CLINICAL TRIAL: NCT04320680
Title: Cohort Follow-up of Systemic Lupus Erythematosus Within the Framework of the Multidisciplinary Consultation at the CHRU of Brest
Brief Title: Systemic Lupus Erythematosus Within the Framework of the Multidisciplinary Consultation
Acronym: CO LUPUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC20.0073
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: cutaneous lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: diagnosis and follow up of a lupus cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lupus cohort follow up (Other): it is a descrption lupus patients study
  Interventions: Other: description of a lupus patient cohort

INTERVENTIONS:
Other: description of a lupus patient cohort — description of a lupus patient cohort

SUMMARY:
Diagnosis and follow up of a lupus cohort in a multidisciplinary consultation in Brest ( France)

DETAILED DESCRIPTION:
all patients coming to the LUPUS multidisciplinary consultation in brest ( France) will have a clinical examination, a biological and immunogical blood samples, cutaneous biopsies or renal biospies if necessary, an ultrasonographic articular and salivary glandular examination if needed. In case of articular involvement, some Xrays ( hands and feet) will be done at the inclusion and during the follow up each year during 5 years .

ELIGIBILITY:
Inclusion Criteria:

* women or men, more than 18 years old, coming to the multidisciplinary consultation in brest ( France).
* With written consentment

Exclusion Criteria:

* patients less than 18 years old
* refusing to participate
* Under legal protection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2025-05-13 (Estimated); Study Completion 2025-05-13 (Estimated)

PRIMARY OUTCOMES:
Cohort lupus: epidemiologic lupus study about diagnosis and follow up | five years
  epidemiologic lupus study in collecting data ( description of the population, biologic and immunologic data collection, data of articular damges with xrays datas) about Diagnosis and follow up of a cohort lupus in a multidisciplibnary consultation in brest hospital ( France).

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement